CLINICAL TRIAL: NCT06141811
Title: A Follow-up Study to Evaluate the Safety of ALLO-ASC-DFU in ALLO-ASC-DFU-302 Clinical Trial
Status: Recruiting | Type: Observational
Sponsor: Anterogen Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: ALLO-ASC-DFU-304
Record Dates: First submitted 2023-11-02; First posted 2023-11-21 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ALLO-ASC-DFU: Subjects with ALLO-ASC-DFU treatment in phase 3 clinical trial of ALLO-ASC-DFU-302
  Interventions: Biological: ALLO-ASC-DFU
- Vehicle sheet: Subjects with Vehicle sheet treatment in phase 3 clinical trial of ALLO-ASC-DFU-302
  Interventions: Procedure: Vehicle sheet

INTERVENTIONS:
Biological: ALLO-ASC-DFU — Application of ALLO-ASC-DFU sheet to Diabetic Foot Ulcer. This study is a follow-up study without intervention.
  Groups: ALLO-ASC-DFU
Procedure: Vehicle sheet — Application of Vehicle sheet to Diabetic Foot Ulcer. This study is a follow-up study without intervention.
  Groups: Vehicle sheet

SUMMARY:
This is a follow-up study to evaluate the safety for the subjects with ALLO-ASC-DFU treatment in phase 3 clinical trial (ALLO-ASC-DFU-302) for 24 months

DETAILED DESCRIPTION:
This is an open-label follow up study to evaluate the safety for the subjects with ALLO-ASC-DFU treatment in phase 3 clinical trial (ALLO-ASC-DFU-302) for 24 months. ALLO-ASC-DFU is a hydrogel sheet containing allogenic adipose-derived mesenchymal stem cells. Adipose-derived stem cells have anti-inflammatory effect and release growth factors such as vascular endothelial growth factor (VEGF) and hepatocyte growth factor (HGF), which can enhance wound healing and regeneration of new tissue, finally may provide a new option in treating a Diabetic Foot Ulcer.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are treated with ALLO-ASC-DFU sheet or Vehicle sheet in phase 3 clinical trial of ALLO-ASC-DFU-302.
2. Subjects who are able to give written informed consent prior to study start and to comply with the study requirements.

Exclusion Criteria:

1. Subjects who are considered not suitable for the study by the principal investigator.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ubjects who are treated with ALLO-ASC-DFU sheet or Vehicle sheet in phase 3 clinical trial of ALLO-ASC-DFU-302.
Sampling Method: Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2023-04-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of systemic tolerance through incidence of abnormal laboratory test results | Up to 9 months
Evaluation of incidence of clinically significant change in physical examination and vital signs | Up to 18 months
Evaluation of localized tolerance through incidence of clinically significant change about treatment area | Up to 24 months
Evaluation of incidence of adverse events | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: ChangSik Park, MD. Ph D, Principal Investigator — Asan Medical Center; JiUng Bak, MD. Ph D, Principal Investigator — Borame Medical Center; DaeWon Jun, MD. Ph D, Principal Investigator — Bucheon St. Mary's Hospital; YoungKoo Lee, MD. Ph D, Principal Investigator — Soonchunhyang University Hospital
Locations (4):
- South Korea (4):
  - Soonchunhyang University Hospital, Bucheon-si, Gyeonggi-do
  - Bucheon ST. Mary's Hospital, Bucheon-si, Gyeonggi-do
  - Asan Medical Center, Seoul
  - Borame Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Undecided